CLINICAL TRIAL: NCT03068780
Title: Double-blind, Randomised, Vehicle-controlled, Phase III, Efficacy and Safety Study With 24-month Open-label Follow-up of Oleogel-S10 in Patients With Inherited Epidermolysis Bullosa
Brief Title: Phase III Efficacy and Safety Study of Oleogel-S10 in Epidermolysis Bullosa
Acronym: EASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amryt Research Limited (Industry)
Responsible Party: Sponsor
Organization: Amryt Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEB-13; 2016-002066-32 (EudraCT Number)
Expanded Access: Available
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — episalvan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oleogel-S10 (Experimental)
  Interventions: Drug: Oleogel-S10
- Control Gel (Placebo Comparator)
  Interventions: Drug: Control gel

INTERVENTIONS:
Drug: Oleogel-S10 — 10% birch bark extract in 90% sunflower oil
  Other Names: Episalvan; Filsuvez
  Arms: Oleogel-S10
Drug: Control gel — Sunflower oil, Cera flava/yellow wax, and Carnauba wax (matched Oleogel-S10 in terms of texture and visual appearance)
  Other Names: Vehicle gel
  Arms: Control Gel

SUMMARY:
This was a Phase III, Efficacy and Safety Study of Oleogel-S10 in Participants with Inherited Epidermolysis Bullosa (EB).

EB is a rare group of genetic skin fragility disorders characterised by blistering of the skin in response to minor injury. In most cases, onset of EB is at birth or shortly after. All participants affected by any type of EB share the main characteristic of repeatedly developing painful wounds that take days to months to heal. Current treatment of EB is primarily preventative and supportive including protection from mechanical forces by avoiding rubbing, early treatment of wounds to prevent infections, and protection of the wound with adequate non-adhesive dressings to enable healing.

The active pharmaceutical ingredient in Oleogel-S10 is a refined birch bark extract, quantified to 72 to 88% betulin.

This clinical study of Oleogel-S10 in patients with inherited EB has been carried out to investigate whether Oleogel-S10 is effective for treatment of EB wounds and safe for long-term use.

Oleogel-S10 was compared to a control gel. The control gel matched Oleogel-S10 in terms of texture and visual appearance to allow for double-blinding. The packaging for Oleogel-S10 gel and the control gel were identical. The participant received either Oleogel-S10 or control gel for a double-blind study phase of 90 days. The probability that the participant received Oleogel-S10 was 50%, which means that they had a 1 in 2 chance of receiving Oleogel-S10. However, in the follow-up phase of the study all participants were treated with Oleogel-S10 for a period of 24 months.

This clinical study was performed at 49 study sites in 26 countries (Argentina, Australia, Austria, Brazil, Chile, Colombia, Czech Republic, Denmark, France, Georgia, Germany, Greece, Hong Kong [China], Hungary, Ireland, Israel, Italy, Romania, Russia, Serbia, Singapore, Spain, Switzerland, Ukraine, United Kingdom, and the United States); 223 participants participated in total.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with the following subtypes of inherited EB: junctional EB (JEB), dystrophic EB (DEB), and Kindler EB aged ≥21 days
* Patients with an EB target wound (i.e., EB partial thickness wound of 10 cm² to 50 cm² in size aged ≥21 days and <9 months)
* Patient and/or his/her legal representative has/have been informed, has/have read and understood the patient information/informed consent form, and has/have given written informed consent
* Patient and/or his/her legal representative must be able and willing to follow study procedures and instructions

Exclusion Criteria:

* Patient has EB simplex
* EB target wound that is ≥9 months old or has clinical signs of local infection
* Use of systemic antibiotics for wound-related infections within 7 days prior to enrolment
* Administration of systemic or topical steroids (except for inhaled, ophthalmic or topical applications, such as budesonide suspension for oesophageal strictures [e.g., Pulmicort respules® 0.25 mg/2 mL or 0.5 mg/2 mL]) within 30 days before enrolment
* Immunosuppressive therapy or cytotoxic chemotherapy within 60 days prior to enrolment
* Patient has undergone stem cell transplant or gene therapy for the treatment of inherited EB
* Current and/or former malignancy including basal cell carcinomas and squamous cell carcinomas
* Enrolment in any interventional study or treated with any investigational drug for any disease within 4 weeks prior to study entry
* Factors present in the patient and/or his/her legal representative that could interfere with study compliance such as inability to attend scheduled study visits or compliance with home dressing changes
* Pregnant or nursing women and women of childbearing potential including postmenarchal female adolescents not willing to use an effective form of birth control with failure rates <1% per year (e.g., implant, injectable, combined oral contraceptive, intrauterine contraceptive device, sexual abstinence, vasectomised partner) during participation in the study (and at least 3 months thereafter)
* Patient is a member of the investigational team or his/her immediate family
* Patient lives in the same household as a study participant

Min Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes S Kern, MD PhD, Principal Investigator — Melbourne Health
Locations (51):
- United States (10):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Colorado, Aurora, Colorado
  - Amjad Plastic Research, Miami, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Stony Brook University Hospital, Stony Brook, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Argentina (3):
  - Consutorios Medicos (Instituto de Neumonologia y Dermatologia), Buenos Aires
  - Centro Médico Dra. De Salvo, Buenos Aires
  - Centro de investigaciones Metabolicas, CINME, Buenos Aires
- Australia (4):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Premier Specialists, Sydney, New South Wales
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Murdoch Childrens Research Institute Royal Children's Hospital, Parkville, Victoria
- Universitaetsklinik fuer Dermatologie, Salzburg, Austria
- Brazil (3):
  - IMIP, Recife, Pernanbuco
  - Universidade Regional de Blumenau, Blumenau, Santa Catarina
  - Instituto Da Crianca HCFMUSP, São Paulo
- Fundacion Debra Chile, Santiago, Chile
- Hospital De San Jose, Bogotá, DC, Colombia
- University Hospital Brno, Children´s Hospital, Brno, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- France (2):
  - Hôpital Necker-Enfants Malades, Paris
  - CHU Toulouse - Hospital Larrey, Toulouse
- S/R National Center of Dermatology and Venerology, Tbilisi, Georgia
- Germany (2):
  - Medical Center University Freiburg, Freiburg im Breisgau
  - Kinder- und Jugendkrankenhaus AUF DER BULT, Hanover
- Hospital of Skin and Veneral Diseases "A. Syggros", Athens, Attica, Greece
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong
- Semmelweis University, Faculty of Medicine, Budapest, Hungary
- Our Ladys Childrens Hospital, Dublin, Ireland
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Bambino Gesù Children Hospital, Roma
  - Istituto Dermopatico dell'Immacolata IDI-IRCCS, Roma
- Centrul Medical Sanador, Bucharest, Romania
- Russia (2):
  - State Scientific Center for Dermatovenerology and Cosmetology, Moscow
  - Scientific Center of Children's Health, Moscow
- University of Belgrade, School of Medicine, Belgrade, Serbia
- Kandang Kerbau (KK) Women's and Children's Hospital, Singapore, Singapore
- Spain (4):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitari de la Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Viamed Santa Ángela de la Cruz, Seville
- Bern University Hospital, Bern, Switzerland
- National Children Specialized Hospital "Ohmatdyt" of Ministry of Health of Ukraine, Kyiv, Ukraine
- United Kingdom (2):
  - Birmingham Children's Hospital NHS Trust, Birmingham
  - Great Ormond Street hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kern JS, Schwieger-Briel A, Lowe S, Sumeray M, Davis C, Martinez AE. Oleogel-S10 Phase 3 study "EASE" for epidermolysis bullosa: study design and rationale. Trials. 2019 Jun 11;20(1):350. doi: 10.1186/s13063-019-3362-z. PMID 31186047

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects satisfied the inclusion / exclusion criteria based on investigator assessment prior to entry into the study. 29 out of a total of 252 screened patients were reported as screen failures.
Groups:
- Oleogel-S10: Oleogel-S10 (DBP & OLP): 10% birch bark extract in 90% sunflower oil
- Control Gel: Control gel (DBP): Vehicle gel; Oleogel-S10 (OLP): 10% birch bark extract in 90% sunflower oil
Period: Double-Blind Phase (DBP)
Arm/Group | Oleogel-S10 | Control Gel
Started | 109 | 114
Completed | 100 | 99
Not Completed | 9 | 15
Period: Open-Label Phase (OLP)
Arm/Group | Oleogel-S10 | Control Gel
Started | 100 | 105 (All subjects switched to Oleogel-S10 in the OLP. 6 subjects, all control gel, discontinued from DBP and entered OLP prematurely.)
Completed | 66 | 75
Not Completed | 34 | 30

BASELINE CHARACTERISTICS:
Groups:
- Control Gel: Control gel: Vehicle gel (all subjects switched to Oleogel-S10 in the OLP)
- Total: Total of all reporting groups
Arm/Group | Oleogel-S10 | Control Gel | Total
Number analyzed (Participants) | 109 | 114 | 223
Age, Customized [Count of Participants; unit: Participants]
  < 4 years | 7 | 10 | 17
  4 to <12 years | 42 | 43 | 85
  12 to <18 years | 25 | 29 | 54
  18 years and older | 35 | 32 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 89
  Male | 68 | 66 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 95 | 91 | 186
  Black or African American | 1 | 2 | 3
  Asian | 4 | 7 | 11
  American Indian or Alaska Native | 0 | 1 | 1
  Unknown | 1 | 1 | 2
  Not applicable (applies in countries where the collection of race was prohibited) | 4 | 8 | 12
  Other (applies if none of the races listed were appropriate or if the subject was of mixed race) | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Europe | 48 | 55 | 103
  South America | 33 | 35 | 68
  United States | 7 | 7 | 14
  Australia | 6 | 2 | 8
  Georgia | 1 | 3 | 4
  Hong Kong | 0 | 2 | 2
  Israel | 9 | 4 | 13
  Russia | 4 | 4 | 8
  Singapore | 1 | 1 | 2
  Ukraine | 0 | 1 | 1
Epidermolysis Bullosa Subtype [Count of Participants; unit: Participants]
  RDEB (recessive dystrophic epidermolysis bullosa) | 91 | 84 | 175
  DDEB (dominant dystrophic epidermolysis bullosa) | 6 | 14 | 20
  JEB (junctional epidermolysis bullosa) | 11 | 15 | 26
  EBS (epidermolysis bullosa simplex) | 1 | 1 | 2
  Kindler EB | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 16.05 (4.979) | 16.31 (5.037) | 16.18 (4.999)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With First Complete Closure of the EB Target Wound Within 45 Days of Treatment
Description: Proportion of subjects with first complete closure of the EB target wound (defined as EB partial-thickness wound of 10 cm2 to 50 cm2 in size and ≥21 days to <9 months in age) in subjects with inherited EB (subtypes DEB, JEB, or Kindler EB) within 45 days of treatment with Oleogel-S10 compared to control gel based on clinical assessment by the investigator (the wound was rated as "closed" at first appearance of complete re-epithelialization without drainage).
Time Frame: 45±7 days
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Groups:
- Control Gel: Control gel: Vehicle gel
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 109 | 114
Participants | 45 | 33
Statistical Analysis 1: Comparison: Oleogel-S10 vs Control Gel; Test type: Superiority; p = 0.013, Cui, Hung, Wang (CHW) approach — P-value adjusted with CHW method using CMH test statistics based on a test stratified by EB subtype and target wound size class estimated separately before and after the interim analysis for sample size re-estimation.Threshold of superiority p<0.05; Primary efficacy endpoint was first assessed with the CMH test, but the final statistical analysis was performed based on the CHW approach; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.02 to 3.30] — The CMH test statistic from the data until the interim analysis (IA) and the CMH test statistic of the data after the IA must be calculated separately. The results are then combined using the CHW weighted approach to one test-statistic

2. Secondary Outcome: Time to First Complete Closure of the EB Target Wound as Evidenced by Clinical Assessment Until Day 90 (D90) or End of Double-blind Phase (EDBP)
Description: The first key secondary endpoint was time to first complete closure of the EB target wound as evidenced by clinical assessment within 90 days or by EDBP, using a nonstratified log-rank test.
  If the primary analysis of the primary efficacy endpoint showed superiority at the 5% significance level, hierarchical confirmatory testing of the 6 key secondary endpoints was to be performed.
Time Frame: 90±7 days
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 109 | 114
days | 92.0 [50 to NA] — Confidence interval for the median time to first complete closure was not estimable since the survivor function of the upper confidence limit did not reach 0.5 (upper limit not estimable) | 94.0 [89 to NA] — Confidence interval for the median time to first complete closure was not estimable since the survivor function of the upper confidence limit did not reach 0.5 (upper limit not estimable)
Statistical Analysis 1: Comparison: Oleogel-S10 vs Control Gel; Test type: Superiority; p = 0.302, Chi-squared — Threshold of superiority is p<0.05

3. Secondary Outcome: Proportion of Patients With First Complete Closure of the EB Target Wound at D90 or EDBP Based on Clinical Assessment by the Investigator Until D90 or EDBP
Description: The second key secondary endpoint was the proportion of subjects with first complete closure of the EB target wound within 90 days of treatment or by EDBP based on clinical assessment by the investigator.
Time Frame: 90±7 days
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 109 | 114
Participants | 55 | 50

4. Secondary Outcome: The Incidence of EB Target Wound Infection Between Baseline (DBP D0) and D90 or EDBP as Evidenced by Adverse Events (AEs) and/or Use of Topical and/or Systemic Antibiotics (Related to Wound Infection)
Description: The incidence of EB target wound infections between Baseline (DBP D0) and D90 or EDBP was assessed based on the total number of patients with an EB target wound infection, as evidenced by AEs and/or the use of topical and/or systemic antibiotics, and the total number of patients
Time Frame: 90±7 days
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 109 | 114
Participants | 1 | 5

5. Secondary Outcome: The Maximum Severity of EB Target Wound Infection Between Baseline (DBP D0) and D90 or EDBP as Evidenced by AEs
Description: Target wound infections between baseline (DBP D0) and D90 or EDBP were assessed for maximum severity (maximum severity was evaluated if a subject had a wound infection event evidenced by AEs). [Note: Here, 1 event less is recorded in the control gel group as for the previous secondary outcome measure, because only wound infections that were reported as AEs could be assessed for severity and were included in this analysis.]
Time Frame: 90±7 days
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 109 | 114
Participants
  Maximum severity of wound infection: Mild | 1 | 0
  Maximum severity of wound infection: Moderate | 0 | 3
  Maximum severity of wound infection: Severe | 0 | 1
  No wound infection | 108 | 110

6. Secondary Outcome: Change From Baseline (DBP D0) in Total Body Wound Burden as Evidenced by Clinical Assessment Using Section I (Assessment of the Skin Except for the Anogenital Region) of the 'EB Disease Activity and Scarring Index' (EBDASI), at D90 or EDBP
Description: The evaluation of total body wound burden (TBWB) was based on clinical assessment using Section I (Skin) of the Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI). The EBDASI skin activity (blistering/erosions/crusting) was scored from 0 to 10 for each of 10 anatomical locations (excluding the anogenital and buttocks regions). Therefore, the total skin activity score (i.e., TBWB) could range from 0 to 100, with lower scores indicative of less wound burden. The change in TBWB was assessed from baseline (DBP D0) to D90 or EDBP.
Time Frame: 90±7 days
Population: Patients with EBDASI skin activity score
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 84 | 85
score on a scale | -0.44 (0.90) | -0.56 (0.85)

7. Secondary Outcome: Change From Baseline (DBP D0) in Itching Using the 'Itch Man Scale' in Patients ≥ 4 Years and up to 13 Years of Age Before Wound Dressing Changes at D90 or EDBP
Description: Change from Baseline at D90 or EDBP on the Itch Man Scale in patients 4-13 years of age. The scale runs from 0 (comfortable, no itch) to 4 (itches most terribly, impossible to sit still, concentrate).
Time Frame: 90±7 days
Population: Patients with Itch Man Score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 39 | 43
score on a scale | -0.44 (1.31) | -1.00 (1.31)

8. Secondary Outcome: Change From Baseline (DBP D0) in Itching Using the 'Leuven Itch Scale' in Patients ≥ 14 Years of Age Before Wound Dressing Changes at D90 or End of Double Blind Phase (EDBP)
Description: Change in Leuven Itch Scale (patients ≥ 14 years of age) scores taken from two time points, Baseline and Day 90±7 [End of Double Blind Phase (EDBP)]. The Leuven Itch Scale measures six dimensions of the itch experience: Frequency Subscore (0 = Never to 100 = Always); Duration Subscore (0 = Between 0 and 30 minutes to 100 = More than 2 hours); Severity Subscore (0 = No itch to 100 = Worst possible itch); Consequences Subscore [0 = Never to 100 = Always (lower score indicates less negative consequences from the itch)]; Distress Subscore (0 = Not distressing at all to 100 = Very distressing); Surface Area Subscore (0-100, high values indicate more parts of the body are itching)
Time Frame: 90±7 days
Population: Patients with Leuven Itch Score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oleogel-S10 | Control Gel
Number analyzed (Participants) | 52 | 48
score on a scale
  Frequency subscore (change from baseline): number analyzed (Participants) | 40 | 37
  Frequency subscore (change from baseline) | -8.13 (26.18) | -10.14 (27.3)
  Duration subscore (change from baseline): number analyzed (Participants) | 36 | 34
  Duration subscore (change from baseline) | -0.93 (35.174) | 0.98 (39.768)
  Severity subscore (change from baseline): number analyzed (Participants) | 36 | 34
  Severity subscore (change from baseline) | -4.95 (19.33) | -10.76 (32.68)
  Consequences subscore (change from baseline): number analyzed (Participants) | 36 | 34
  Consequences subscore (change from baseline) | -4.39 (14.073) | -3.54 (19.402)
  Distress subscore (change from baseline): number analyzed (Participants) | 35 | 34
  Distress subscore (change from baseline) | -0.44 (22.87) | -0.26 (34.87)
  Surface area subscore (change from baseline): number analyzed (Participants) | 35 | 34
  Surface area subscore (change from baseline) | -1.54 (12.347) | 0.68 (17.082)

ADVERSE EVENTS:
Time Frame: DBP D0 to the last dose of study medication at Month 24 (OLP) ±14 days
Groups:
- Oleogel-S10 (DBP); Former Oleogel-S10 (OLP); Former Control Gel (OLP): Oleogel-S10: 10% birch bark extract in 90% sunflower oil
- Control Gel (DBP): Control gel: Vehicle Gel
Arm/Group | Oleogel-S10 (DBP) | Control Gel (DBP) | Former Oleogel-S10 (OLP) | Former Control Gel (OLP)
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/114 | 7/100 | 2/105
Serious Adverse Events (participants affected / at risk) | 7/109 | 6/114 | 26/100 | 24/105
Other Adverse Events (participants affected / at risk) | 89/109 | 92/114 | 77/100 | 81/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oleogel-S10 (DBP) (N=109) | Control Gel (DBP) (N=114) | Former Oleogel-S10 (OLP) (N=100) | Former Control Gel (OLP) (N=105)
septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (9) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 4 (7) | 6 (8)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pseudosyndactyly (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia/ (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection bacterial (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syndactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemmorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Ischemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal mucosal blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic congestion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oleogel-S10 (DBP) (N=109) | Control Gel (DBP) (N=114) | Former Oleogel-S10 (OLP) (N=100) | Former Control Gel (OLP) (N=105)
Wound complication (Injury, poisoning and procedural complications) | 67 (100) | 61 (88) | 38 (43) | 46 (64) — Refers to any AEs under PT "wound complication." These include increase in wound size vs. baseline or previous visit, wound reopening, wound injury, increase in wound burden, worsening of EB wound pain, wound odor, and wound worsening vs baseline.
Wound infection (Infections and infestations) | 8 (9) | 10 (12) | 6 (12) | 15 (26)
Wound infection staphylococcal (Infections and infestations) | 4 (4) | 3 (3) | 9 (14) | 12 (15)
Wound infection bacterial (Infections and infestations) | 3 (4) | 5 (6) | 7 (10) | 9 (14)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 8 (16) | 11 (14)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (8) | 7 (9)
Anaemia (Blood and lymphatic system disorders) | 8 (10) | 4 (4) | 16 (24) | 21 (30)
Pyrexia (General disorders) | 9 (11) | 15 (18) | 10 (13) | 10 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (7) | 5 (5) | 9 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (9) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 6 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 5 (8) | 5 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7) | 3 (3) | 1 (2)
Influenza (Infections and infestations) | 2 (2) | 6 (6) | 1 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT03068780/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT03068780/SAP_001.pdf